CLINICAL TRIAL: NCT00613158
Title: Atherosclerosis Risk Refinement - a Multi-marker Approach Using Microarrays
Brief Title: Using Differences in Peripheral Blood Leukocyte Gene Expression to Determine Cardiovascular Disease Risk
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Chiang-Ching Huang, PhD, Northwestern University
Other Study IDs: 1384; R01HL086678-01A1 (NIH)
Record Dates: First submitted 2008-02-08; First posted 2008-02-12 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-04

CONDITIONS: Atherosclerosis; Cardiovascular Diseases
Keywords: Subclincal Atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Participants from the Multi-Ethnic Study of Atherosclerosis (MESA) with significant subclinical atherosclerosis (SA) and a low Framingham risk score
- 2: Participants from MESA with no SA and a low Framingham risk score
- 3: Healthy participants from Northwestern University

SUMMARY:
Cardiovascular disease (CVD), including heart disease, heart attack, high blood pressure, and stroke, is most commonly caused by atherosclerosis, or a hardening of the arteries. Traditional risk factors for CVD include age, high blood pressure, high cholesterol, diabetes, and smoking. Although these established risk factors can be helpful in determining people at risk for developing CVD, the addition of novel gene markers for subclinical, or suspected, atherosclerosis (SA) may enhance CVD risk prediction and understanding of disease mechanisms. This study will compare specific genes of white blood cells in people with significant SA versus people without SA to improve identification of those at risk for developing CVD and to better understand the biological basis of SA.

DETAILED DESCRIPTION:
CVD is the leading cause of death worldwide and accounts for almost 40% of deaths each year in the United States. In a person with CVD, oxygenated blood is not adequately distributed throughout the body because of impaired function in the heart and blood vessels. This restricted blood flow can eventually lead to organ damage, heart attack, and stroke. Risk prediction for CVD, which is largely associated with SA, relies on the use of certain traditional risk factors. The widely used Framingham risk score (FRS) has provided excellent risk discrimination and reliable estimates of 10-year risk for CVD, but it does not account for the genetics behind SA. Although numerous studies have investigated novel genetic biomarkers to attempt to add predictive value to the FRS, no single biomarker to date has been able to improve risk prediction in a meaningful way. A multi-marker approach that identifies several novel markers unrelated to traditional risk factors may be more effective in improving the identification of those at risk for CVD. This study will first construct a multi-marker approach that is based on patterns of gene expression in peripheral blood leukocytes (PBLs) and that can serve to identify people with substantial SA. The study will then use this approach to determine whether gene expression patterns of PBLs in people with SA are distinct from those in people without SA.

This study will use previously collected data and specimens, including blood samples and SA imaging, from participants in the Multi-Ethnic Study of Atherosclerosis (MESA) trial and from healthy female participants from Northwestern University. Blood samples will be used for analysis of patterns of gene expression in PBLs. There will be no new study visits for this study.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Inclusion Criteria:

* Female participant from the MESA study who has a low Framingham risk score and has either SA or no evidence of SA
* Healthy female below the age of 40 from Northwestern University.

Exclusion Criteria:

- Diabetes

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include female participants from MESA with and without SA. This study will also include healthy female participants from Northwestern University.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-03; Primary Completion 2007-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
SA burden, as indicated by coronary artery calcium score and intima-medial thickness | Measured at completion of sample analysis

CONTACTS AND LOCATIONS:
Overall Officials: Chiang-Ching Huang, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States